CLINICAL TRIAL: NCT04818281
Title: Phase I Study Evaluating the Basic Pharmacological and Toxicological Effects of the Protective VLP Vaccine Developed Against SARS-CoV-2 in Healthy Participants, Administered as Two Injections Subcutaneously, in Two Different Dosages.
Brief Title: Study of a Severe Acute Respiratory Syndrome CoV-2 (SARS-CoV-2) Virus-like Particle (VLP) Vaccine in Healthy Adults
Acronym: COVID-19
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ihsan GURSEL, PhD, Prof. (Other)
Collaborators: Dr Abdurrahman Yurtaslan Ankara Oncology Training and Research Hospital (Other); The Scientific and Technological Research Council of Turkey (Other); MonitorCRO (Industry); Nobel Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Ihsan GURSEL, PhD, Prof., PhD, Prof, The Scientific and Technological Research Council of Turkey
Organization: The Scientific and Technological Research Council of Turkey (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VLP-58-1023-Al-K3
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Covid19
Keywords: Virus-like Particles harboring S, M, N, E antigens; SARS-CoV-2; K3-CpG ODN; Alum
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Dose Group (Group A) (Experimental): 12 participants will receive 10 µg VLP vaccine (adjuvanted with alum and CpGODN-K3)
  Interventions: Biological: SARS-CoV-2 VLP Vaccine
- High-Dose Group (Group B) (Experimental): 12 participants will receive 40 µg VLP vaccine (adjuvanted with alum and CpGODN-K3)
  Interventions: Biological: SARS-CoV-2 VLP Vaccine
- Placebo Group (Placebo Comparator): 12 participants will receive 1 ml of 0.9% sodium chloride (NaCl)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: SARS-CoV-2 VLP Vaccine — VLP adjuvanted vaccine
  Arms: High-Dose Group (Group B); Low-Dose Group (Group A)
Biological: Placebo — 0.9% NaCl
  Arms: Placebo Group

SUMMARY:
This is a VLP SARS-CoV-2 vaccine study of a vaccine developed in Turkey and manufactured according to Good Manufacturing Practices (GMP) requirements. Preclinical toxicology studies on experimental animals are to be concluded. The purpose of this Phase I study is to examine the safety, tolerability, and immunogenicity of the protective VLP vaccine against SARS-CoV-2, which will be administered by a double-blind, randomized method, in two different doses (low dose and high dose).

DETAILED DESCRIPTION:
This phase I study is designed as double-blinded, randomised, placebo controlled, three-armed study composed of two different dose arms of protective VLP vaccine (harboring M, N, E, and hexapro modified S proteins of SARS-CoV-2 virus) against SARS-CoV-2 in dose escalations (first low dose group, followed by high dose group) and placebo arm. Each dose of vaccine will be defined as a cohort in itself, with vaccine administration to 12 participants and placebo administration to 6 participants. After completion of low-dose group, decision of switch to high-dose will be taken by the Independent Data Monitoring Committee and study will continue accordingly.

The study will be completed in 12 months.

All injections will be done subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for the study, each participant must satisfy all the following criteria:

1. Healthy participants between 18-59 years of age,
2. Sign an informed consent document,
3. Negative immunoglobulin G (IgG) and immunoglobulin M (IgM) antibody for COVID-19,
4. Negative quantitative polymerase chain reaction (qPCR) SARS-CoV-2 results of nasopharyngeal/sputum samples,
5. Able to comply with the study protocol during the study period,
6. Negative tests for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV),
7. Body temperature <37.2 C,
8. Body mass index 18-35 kg/m2,
9. Normal laboratory levels of whole blood count, alanine transaminase (ALT), aspartate transaminase (AST), total bilirubin, urea, creatinine, and fasting blood glucose,
10. Good general health (no known disease in the history and physical examination within 14 days prior to the enrolment),
11. Female participants who are not pregnant or who will be able to have appropriate contraception methods within 30 days prior to vaccine injection and within 6 months after vaccination,
12. Male participants who will be able to have appropriate contraception methods for 6 months after vaccination,

Exclusion Criteria:

Participants with any of the following criteria will be excluded:

1. History of seizure, encephalopathy or psychosis,
2. History of allergic reactions to any known vaccine or to any component of the study vaccine,
3. Pregnant, breastfeeding or positive pregnancy test or planning to conceive within 6 months,
4. Active infection signs or body temperature >37.2 C,
5. History of SARS-CoV-2 infection,
6. Severe cardiovascular disorders (arrhythmia, conduction disorders, history of myocardial infarction, uncontrolled hypertension),
7. Severe chronic disorders (asthma, diabetes mellitus, thyroid disorders…etc),
8. Congenital or acquired angioedema,
9. Diagnosis of immunodeficiency,
10. Diagnosis of bleeding diathesis,
11. Use of immunosuppressive treatment, anti-allergic treatment, cytotoxic treatment, inhaler corticosteroids (allergic rhinitis or topical steroid ointments are excluded),
12. Those who received blood and blood product transfusions in the last 6 months,
13. Those on any vaccine program or experimental medication within 1 month prior to the study,
14. History of any live vaccine administration within 1 month prior to the study,
15. History of any inactive vaccine administration within 1 month prior to the study,
16. Use of active tuberculosis treatment,
17. According to the investigator's evaluation, those who have any condition (medical, psychological, social, etc.) that may impair the patient's compliance with the study will be excluded from the study.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2021-03-27 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Acute adverse events (AEs) | 24 hours
  Frequency of acute AEs in all dosage groups
Solicited local and systemic adverse events (AEs) | 6 days
  Frequency of local and systemic AEs in all dosage groups
Unsolicited local and systemic adverse events (AEs) | 28 days
  Frequency of local and systemic AEs in all dosage groups

SECONDARY OUTCOMES:
Specific antibody (IgG) response | Before booster dose administration, on Day 14-21-28 and at the end of Month 3 and Month 6 after booster dose
  IgG type antibody titers against anti-Spike protein of SARS-CoV-2 (by ELISA)
Neutralizing antibody response | Before booster dose administration, on Day 14-21-28 and at the end of Month 3 and Month 6 after booster dose
  Neutralizing antibody titer against anti-Spike protein by virus neutralization method developed against SARS-CoV-2
Cellular immune response (IL-4) | Before booster dose administration, on Day 14-21-28 and at the end of Month 3 and Month 6 after booster dose
  ELISPOT: Interleukin-4 (IL4) positive cell level of peripheral blood mononuclear cells (PBMCs) stimulated with rec. S protein
Cellular immune response (IFN-γ) | Before booster dose administration, on Day 14-21-28 and at the end of Month 3 and Month 6 after booster dose
  ELISPOT: Interferon-γ (IFN-γ) positive cell level of peripheral blood mononuclear cells (PBMCs) stimulated with rec. S protein

CONTACTS AND LOCATIONS:
Locations (1):
- Dr. Abdurahman Yurtaslan Ankara Oncology Training and Research Hospital Phase I Clinical Study Center, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Yilmaz IC, Ipekoglu EM, Golcuklu BS, Bildik T, Aksoy AGB, Evcili I, Turay N, Surucu N, Bulbul A, Guvencli N, Yildirim M, Canavar Yildirim T, Atalay YA, Abras I, Ceylan Y, Ozsurekci Y, Tigen ET, Korten V, Gursel M, Gursel I. A phase I/II study of CpG/alum-adjuvanted mammalian-derived quadruple antigen carrying virus-like particle COVID-19 vaccine. Vaccine. 2025 Mar 7;49:126787. doi: 10.1016/j.vaccine.2025.126787. Epub 2025 Jan 31. PMID 39892108